CLINICAL TRIAL: NCT04014998
Title: Investigation of the Effectiveness of Virtual Reality Applications in Addition to Exercise Program in People With Chronic Neck Pain
Brief Title: Effectiveness of Virtual Reality in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Research Assisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR2805
Record Dates: First submitted 2019-07-05; First posted 2019-07-10 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pain, Neck; Virtual Reality; Proprioception; Balance
Keywords: neck pain; virtual reality; proprioception; balance
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Virtual Reality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual Reality + Exercise
  Interventions: Other: Virtual Reality
- Exercise (Other): Exercise Only
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Virtual reality group will have virtual reality for 20 minutes in addition to motor control exercises for 20 minutes. Virtual reality will apply using Oculus Go. On the other hand control group will have only exercise for 40 minutes. Exercises will include same exercises in both groups, but exercise group will perform exercises twice compared to virtual reality group.
  Other Names: Exercise

SUMMARY:
Virtual reality application has been increasing in recent years for pain control, distraction in wound care, treatment of anxiety disorders and support for physical rehabilitation. For example, it has been found to be effective in reducing pain when used in addition to medical treatment during bandaging of severe burns. The studies related with chronic pain patients were stated that virtual reality application was found to be interactive and fun by patients. Therefore, The aim of this study was to investigate the effects of virtual reality on pain threshold, disability, balance, proprioception, exercise sustainability, muscular performance in neck region, quality of life and anxiety / depression in addition to the exercise program that includes stabilization exercises in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* to have pain more than 3 months,
* to be sedentary,
* to have Neck Disability Index score more than 10.

Exclusion Criteria:

* to have neurological deficits, vestibular pathology, history of surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Joint position sense error will assessed by Cervical Range of Motion device. | Change from baseline joint position sense error (cervical flexion, extension, lateral flexions and rotations) after 6 weeks.
  Joint position sense error will assessed by Cervical Range of Motion device.
Balance will assessed by Dynamic Posturography. | Change from baseline sensorial organization test (vestibular, visual and proprioceptive components), limits of stability (reaction time, movement velocity, endpoint excursion, maximum excursion, directional control) and unilateral stance after 6 weeks.
  Balance will assessed by Dynamic Posturography.

SECONDARY OUTCOMES:
cervical lordosis angle | Change from baseline cervical lordosis after 6 weeks.
  Angle will measure using the plane of the superior vertebral plateau of C7 vertebra and of the inferior plateau of C2.
Kinesiophobia will assessed by Tampa kinesiophobia Scale | Change from baseline kinesiophobia after 6 weeks.
  Kinesiophobia will assessed by Tampa kinesiophobia Scale
Quality of life will assessed by Short-form 36. | Change from baseline quality of life after 6 weeks.
  Quality of life will assessed by Short-form 36.
Disability will assessed by Profile Fitness Mapping Questionnaire(Turkish). | Change from baseline disability after 6 weeks.
  Disability will assessed by Profile Fitness Mapping Questionnaire(Turkish).
Anxiety-depression will assessed by Hospital Anxiety-depression scale. | Change from baseline anxiety-depression after 6 weeks.
  Anxiety-depression will assessed by Hospital Anxiety-depression scale.
Shoulder protraction and forward head posture were assessed by photography method. | Change from baseline shoulder protraction and forward head posture after 6 weeks.
  Shoulder protraction and forward head posture were assessed by photography method.
Pain threshold will assessed by algometer device. | Change from baseline pain threshold of both the right and left upper trapezius, the right and left articular pillar between cervical 1 and 2, the right and left cervical 5 and 6 after 6 weeks.
  Pain threshold will assessed by algometer device.
Pain intensity will assessed with Visual Analog Scale. | Change from baseline pain intensity after 6 weeks.
  Pain intensity will assessed with Visual Analog Scale.
muscle strength will assessed by dynamometer and biofeedback device | Change from baseline muscle strength after 6 weeks.
  muscle strength will assessed by dynamometer and biofeedback device

CONTACTS AND LOCATIONS:
Overall Officials: Halil Kamil Öge, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307